CLINICAL TRIAL: NCT00024440
Title: Randomized Study Of Fludarabine And Cyclophosphamide With Or Without Genasense (Bcl-2 Antisense Oligonucleotide) In Subjects With Relapsed Or Refractory Chronic Lymphocytic Leukemia
Brief Title: Fludarabine and Cyclophosphamide With or Without Oblimersen in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068932; GENTA-GL303; UCLA-0104008
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-10

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; oblimersen; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: filgrastim
Biological: oblimersen sodium
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Oblimersen may help fludarabine and cyclophosphamide kill more cancer cells by making them more sensitive to the drugs. It is not yet known if fludarabine and cyclophosphamide are more effective with or without oblimersen.

PURPOSE: Randomized phase III trial to compare the effectiveness of fludarabine and cyclophosphamide with or without oblimersen in treating patients who have relapsed or refractory chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the complete response and nodular partial response of patients with relapsed or refractory chronic lymphocytic leukemia treated with fludarabine and cyclophosphamide with or without oblimersen.
* Compare the overall response rate, response duration, survival, and time to progression in patients treated with these regimens.
* Compare the clinical benefit and safety of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to disease response to prior fludarabine-containing therapy (responsive vs refractory), number of prior regimens (1-2 vs 3 or more), and duration of response to last prior therapy (more than 6 months vs 6 months or fewer). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oblimersen IV continuously on days 1-7 via an infusion pump (ending on day 8) and fludarabine IV over 20-30 minutes and cyclophosphamide IV over 30-60 minutes on days 5-7. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 11 and continuing until blood counts recover.
* Arm II: Patients receive fludarabine IV over 20-30 minutes followed by cyclophosphamide IV over 30-60 minutes on days 1-3. Patients also receive G-CSF SC beginning on day 7 and continuing until blood counts recover.

Treatment in both arms continues every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month and then every 2 months for 2 years.

PROJECTED ACCRUAL: A total of 200 patients (100 per arm) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed or refractory chronic lymphocytic leukemia (CLL) requiring therapy

  * Primary resistance, defined as disease progression without response during at least 2 courses of myelosuppressive therapy OR
  * Relapsed disease, defined as a response (remission or plateau) followed by relapse on or off prior therapy
  * At least 1 prior regimen must have contained fludarabine
* Intermediate or high-risk CLL

  * Intermediate-risk disease must satisfy at least 1 of the following criteria for active disease:

    * Massive or progressive splenomegaly and/or lymphadenopathy

      * Spleen tip greater than 6 cm below costal margin
    * More than 10% weight loss within the past 6 months
    * Grade 2 or 3 fatigue
    * Fevers greater than 100.5 degrees F or night sweats for more than 2 weeks without evidence of infection
    * Progressive lymphocytosis with an increase of more than 50% over a 2-month period or an anticipated doubling time of less than 6 months
    * Worsening anemia or thrombocytopenia
* Measurable disease with all of the following:

  * Absolute lymphocytosis greater than 5,000/mm^3
  * Lymphocytosis of small to moderate-size lymphocytes with less than 55% prolymphocytes, atypical lymphocytes, or lymphoblasts morphologically determined by manual differential
  * Bone marrow aspirate smear with at least 30% nucleated cells that are lymphoid or a bone marrow core biopsy showing lymphoid infiltrates compatible with CLL
  * Normocellular or hypercellular bone marrow
  * Lymphocyte immunophenotype that shows a predominant B-cell monoclonal population
* No Rai stage 0 CLL or stable CLL not requiring therapy
* No secondary leukemia or history of antecedent hematologic disorder prior to initial onset of CLL (e.g., myelodysplasia)

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Platelet count at least 50,000/mm^3 (hematopoietic growth factor or transfusion independent)
* Negative Coombs' test
* No bleeding or coagulation disorder
* No history of hemolytic anemia, including autoimmune hemolytic anemia
* No history of autoimmune thrombocytopenia

Hepatic:

* Albumin at least 3.0 g/dL
* Bilirubin no greater than 2 mg/dL
* AST no greater than 1.5 times upper limit of normal (ULN) (5 times ULN if due to CLL)
* PT no greater than 1.5 times ULN OR
* INR no greater than 1.3
* PTT no greater than 1.5 times ULN
* No chronic hepatitis or cirrhosis

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No uncontrolled congestive heart failure
* No active symptoms of coronary artery disease (i.e., uncontrolled arrhythmia or recurrent chest pain despite prophylactic medication)
* No New York Heart Association class III or IV disease
* No cardiovascular signs or symptoms grade 2 or greater

Other:

* Able to maintain an ambulatory infusion pump
* HIV negative
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No known hypersensitivity to phosphorothioate-containing oligonucleotides, fludarabine, or cyclophosphamide
* No concurrent medical disease that would preclude study participation
* No uncontrolled seizure disorder
* No unresolved serious infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior autologous or allogeneic stem cell transplantation
* At least 3 weeks since prior immunologic therapy, cytokine therapy, vaccine therapy, or other biologic therapy for CLL and recovered
* No concurrent interleukin-11

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy:

* No concurrent corticosteroid therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy for CLL and recovered

Surgery:

* No prior organ allograft
* At least 3 weeks since prior major surgery for CLL and recovered

Other:

* At least 3 weeks since other prior therapy for CLL and recovered
* No other concurrent investigational therapy
* No concurrent therapeutic anticoagulation
* No concurrent immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley R. Frankel, MD, Study Chair — Genta Incorporated
Locations (1):
- Genta Incorporated, Berkeley Heights, New Jersey, United States

REFERENCES:
- [Result] O'Brien S, Moore JO, Boyd TE, Larratt LM, Skotnicki AB, Koziner B, Chanan-Khan AA, Seymour JF, Gribben J, Itri LM, Rai KR. 5-year survival in patients with relapsed or refractory chronic lymphocytic leukemia in a randomized, phase III trial of fludarabine plus cyclophosphamide with or without oblimersen. J Clin Oncol. 2009 Nov 1;27(31):5208-12. doi: 10.1200/JCO.2009.22.5748. Epub 2009 Sep 8. PMID 19738118
- [Result] O'Brien S, Moore JO, Boyd TE, Larratt LM, Skotnicki A, Koziner B, Chanan-Khan AA, Seymour JF, Bociek RG, Pavletic S, Rai KR. Randomized phase III trial of fludarabine plus cyclophosphamide with or without oblimersen sodium (Bcl-2 antisense) in patients with relapsed or refractory chronic lymphocytic leukemia. J Clin Oncol. 2007 Mar 20;25(9):1114-20. doi: 10.1200/JCO.2006.07.1191. Epub 2007 Feb 12. PMID 17296974